CLINICAL TRIAL: NCT02001181
Title: A Phase 2a, Multi-site, Randomized, Double-blind, Vehicle-controlled, Parallel-group Study Of The Pilot Efficacy, Safety, Tolerability, And Pharmacokinetics Of 2% Tofacitinib Ointment In Subjects With Mild To Moderate Atopic Dermatitis
Brief Title: Tofacitinib Ointment For Atopic Dermatitis (Atopic Eczema)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921214
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; Atopic Eczema; Eczema; topical treatment; skin diseases; tofacitinib; CP-690; 550; Janus Kinase inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: Tofacitinib ointment 20mg/g
- Treatment B (Placebo Comparator)
  Interventions: Drug: Placebo ointment (Vehicle)

INTERVENTIONS:
Drug: Tofacitinib ointment 20mg/g — Tofacitinib ointment 20mg/g twice daily (BID) for 4 weeks
  Arms: Treatment group A
Drug: Placebo ointment (Vehicle) — Placebo ointment (vehicle) twice daily (BID) for 4 weeks
  Arms: Treatment B

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of 2% tofacitinib ointment (20 mg/g) BID (twice daily) in subjects with mild to moderate atopic dermatitis compared to placebo (vehicle) BID for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of atopic dermatitis (also known as atopic eczema) for at least 6 months prior to Day 1 that has been clinically stable for at least 1 month prior to Day 1 and is confirmed to be atopic dermatitis according to the criteria of Hanifin and Rajka.
* Have a PGA score of 2 (mild) or 3 (moderate) at Day 1.
* Have atopic dermatitis on the head (including face, but excluding hair bearing scalp), neck, trunk (excluding groin and genitals), or limbs including palms and soles covering at least 2% of total body surface area (BSA) and up to and including 20% of total BSA at Day 1. At least 2% of the total BSA will need to be on the head (including face, but excluding hair bearing scalp), neck, trunk (excluding groin and genitals), or limbs (excluding palms and soles).

Exclusion Criteria:

* Evidence of certain skin conditions/infections at baseline
* Currently have atopic dermatitis on groin, genitals, palm or soles
* Have certain laboratory abnormalities at baseline
* Females who are pregnant, breastfeeding, or are of childbearing potential not using highly effective contraception

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Canada (5):
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec

REFERENCES:
- [Derived] Purohit VS, Ports WC, Wang C, Riley S. Systemic Tofacitinib Concentrations in Adult Patients With Atopic Dermatitis Treated With 2% Tofacitinib Ointment and Application to Pediatric Study Planning. J Clin Pharmacol. 2019 Jun;59(6):811-820. doi: 10.1002/jcph.1360. Epub 2018 Dec 17. PMID 30556911
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921214&StudyName=Tofacitinib%20Ointment%20For%20Atopic%20Dermatitis%20%28Atopic%20Eczema%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility included male or female participants, 18 to 60 years of age (inclusive), who had a clinical diagnosis of atopic dermatitis for at least 6 months and clinically stable for >=1 month.
Pre-assignment Details: During the screening/washout period, participants' current therapies (topical, systemic, and phototherapy) for atopic dermatitis were discontinued and only non-medicated study emollient, sunscreen topical products, and specific shampoos (for atopic dermatitis on hair-bearing scalp) were permitted.
Groups:
- Tofacitinib 20 mg/g BID: Participants received tofacitinib (20 milligrams per gram [mg/g, 2%]) topical ointment to the treatment area twice a day (BID) for 4 weeks.
- Vehicle BID: Participants received placebo topical ointment vehicle to the treatment area BID for 4 weeks.
Period: Overall Study
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Started | 35 | 34
Completed | 34 | 31
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (9.8) | 30.4 (10.4) | 31.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 4
Description: The EASI quantifies the severity of a participant's atopic dermatitis based on both lesion severity and the percent of BSA affected. The EASI is a composite scoring by the atopic dermatitis clinical evaluator of the degree of erythema, induration/papulation, excoriation, and lichenification (each scored separately) for each of 4 body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of atopic dermatitis. What is reported is the percent change from baseline in EASI scores.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: The full analysis set (FAS) included all participants who were randomized and received at least 1 dose of study drug. Missing data was not imputed. N=number of participants who were in FAS and had a baseline value and an observation at Week 4.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Number analyzed (Participants) | 34 | 31
percent change | -81.7 (6.31) | -29.9 (6.46)
Statistical Analysis 1: Comparison: Tofacitinib 20 mg/g BID vs Vehicle BID; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The mixed model for repeated measures analysis included all the participants in FAS; Mean Difference (Final Values) = -51.8, 80% CI 2-sided [-62.8 to -40.8], Standard Error of Mean 8.48

2. Secondary Outcome: Proportion of Participants Achieving Physician's Global Assessment (PGA) Response of Clear or Almost Clear at Week 4
Description: The PGA score assesses the overall severity of atopic dermatitis. Scores range from 0 to 4 and correspond to a category (clear, almost clear, mild, moderate, and severe, respectively) based on morphological descriptors.
Time Frame: Week 4
Population: The FAS included all participants who were randomized and received at least 1 dose of study drug. Participants who were in FAS and had a baseline PGA score of 2 or 3 were included in the analysis. Participants with missing data at Week 4 were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Number analyzed (Participants) | 35 | 34
percentage of participants | 71.4 | 20.6

3. Secondary Outcome: Proportion of Participants With Response of Clear or Almost Clear and Greater Than or Equal to (>=) 2 Grade/Point Improvement From Baseline at Week 4
Description: as for outcome 2
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Number analyzed (Participants) | 35 | 34
percentage of participants | 65.7 | 11.8

4. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) Efficacy at Week 4
Description: The percent BSA with atopic dermatitis in a body region was determined by the number of handprints of atopic dermatitis skin in that region: head and neck, upper limbs, trunk including axillae, lower limbs including buttocks. In the handprint method, the full palmar hand of the participant (i.e., the participant's fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. What is reported is the percent change from baseline in BSA affected.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: The FAS included all participants who were randomized and received at least 1 dose of study drug. Missing data was not imputed. N=number of participants who were in FAS and had a baseline value and an observation at Week 4.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Number analyzed (Participants) | 34 | 31
percent change | -72.7 (34.1) | -30.2 (39.4)

5. Secondary Outcome: Change From Baseline in the EASI Clinical Signs Severity Sum Score at Week 4
Description: The EASI Clinical Signs Severity Sum Score was derived from the EASI. The Clinical Signs Severity Scores on the 4-point scale for dermatitis lesions were summed in each EASI body region. The sum of the Clinical Signs Severity Score in each EASI body region was then totaled across the 4 EASI body regions to provide an EASI Clinical Signs Severity Sum Score, which ranged from 0 to 48, with higher scores representing greater severity of atopic dermatitis.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Number analyzed (Participants) | 34 | 31
units on a scale | -11.4 (5.3) | -4.1 (4.5)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tofacitinib 20 mg/g BID | Vehicle BID
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 11/35 | 19/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 20 mg/g BID (N=35) | Vehicle BID (N=34)
Conjunctivitis allergic (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Application site pain (General disorders) | 1 | 0
Application site pruritus (General disorders) | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Initial insomnia (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.